CLINICAL TRIAL: NCT00189592
Title: Plantar Fasciosis Treatment Using Coblation® Prospective, Double-Blind, Randomized Controlled Study
Brief Title: Plantar Fasciosis Treatment Using Coblation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ArthroCare Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0105WW
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Plantar Fasciitis
Keywords: plantar fascia; plantar fasciitis; Coblation; fasciotomy; conventional surgical fasciotomy; heel spur; heel pain; aponeurosis; plasma based radiofrequency; angiogenesis
MeSH Terms: conditions — Fasciitis, Plantar; Heel Spur

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Percutaneous Fasciotomy
  Interventions: Device: ArthroCare TOPAZ™ MicroDebrider™ using Coblation
- 2 (Active Comparator): Standard Fasciotomy
  Interventions: Procedure: Surgical Fasciotomy

INTERVENTIONS:
Device: ArthroCare TOPAZ™ MicroDebrider™ using Coblation — Percutaneous treatment of plantar fascia using the Topaz device. No incision performed.
  Arms: A
Procedure: Surgical Fasciotomy — Standard surgical fasciotomy using an incision to treat the plantar fascia.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Coblation-based fasciotomy for relieving pain associated with recurring plantar fasciosis and, secondarily, to determine whether there may be additional potential benefits stemming from its use.

DETAILED DESCRIPTION:
Severe recalcitrant heel pain, resulting from repetitive trauma to the plantar fascia, is a relatively commonly observed phenomenon. Although this condition is frequently referred to as 'heel spurs', plantar fasciitis (acute inflammatory stage) and plantar fasciosis (chronic degeneration) are currently accepted as the more accurate terms. Symptoms most often occur during the first few steps in the morning but may also be effected during intense activity or with prolonged standing. The source of pain symptoms, which are usually perceived as a gradual onset of burning, is located at the origin of the plantar fascia at the calcaneous (heel bone). Risk factors such as low or high arches or over-pronation of the foot, systemic disease, or obesity may exacerbate pain.

More than two million Americans receive treatment each year for plantar fasciitis and fasciosis. Conservative treatment options for plantar fasciosis include rest, stretching, strengthening, and massage, progressing to non-steroidal anti-inflammatories, steroid injections or iontophoresis with continued recalcitrance. Orthotics, heel cups, night splints and plantar strapping are other conservative options frequently recommended by treating physicians. Patient outcomes and response to conservative measures are usually positive, with non-responsive cases, approximately 10% of all presenting cases, receiving surgical care. Extracorporeal shockwave treatment has recently been advocated for the recalcitrant cases and has shown to be effective in 60-80 percent of the cases. Plantar fascia release, either partial or complete, is commonly the surgical procedure of choice for treating plantar fasciosis. However, this surgery has a risk of complications and is thought to alter the biomechanics of the foot, which may be linked to post-operative lateral column pain and long-term disability. Because of the potential postoperative sequelae with plantar fascia release, it is valuable to examine less invasive surgical techniques for treating recalcitrant plantar fasciosis.

The concept of using a plasma RF-based microsurgical approach as a viable modality for treating tendinosis, and now, recalcitrant plantar fasciosis, was originally drawn from the research work conducted in patients treated for congestive heart failure using laser or RF-based transmyocardial revascularization (TMR). The mechanism of action behind the clinical success observed with laser and RF-based TMR was theorized to be associated with the localized angiogenic healing response noted to occur following the procedure. Localized angiogenesis had not been observed previously using mechanical devices for TMR, which were also less successful clinically. To substantiate adopting a TMR-like approach for treating tendinosis, the capability of plasma RF-based microsurgery for initiating an angiogenic healing response was examined in vivo using histology and biochemical analysis. The sum of several studies provides good evidence to suggest that plasma RF-based microsurgery can promote an angiogenic healing response using an appropriate application.

Preliminary clinical experience following plasma RF-based micro-tenotomy has demonstrated excellent success in treating chronic, refractive tendinosis. The investigators reported that this technique was technically simple to perform and was much less invasive than conventional surgery. Patients had a rapid and uncomplicated recovery and reported minimal to no pain 7-10 days following the procedure; their pain relief persisted or improved through 24 months. Magnetic resonance imaging correlated well with clinical results. These promising clinical findings, as well as the evidence from the basic research studies, led us to consider evaluating this plasma RF-based approach for treating symptomatic, chronic, recalcitrant heel pain resembling plantar fasciosis. The purpose of this study is to evaluate the effectiveness of Coblation-based fasciotomy for relieving pain associated with recalcitrant plantar fasciosis and, secondarily, to determine whether there may be additional potential benefits stemming from its use, such as reduced incidence of postoperative complications and improved function, compared to conventional surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plantar fasciitis/fasciosis by all of the following:

  * Tenderness with palpation and local pressure over the medial calcaneal tuberosity on passive dorsiflexion of the foot
  * VAS (Visual Analog Scale) pain score of > 5 points on a scale of 0 to 10, during the first few minutes of walking in the morning
  * Ultrasound or magnetic resonance imaging (MRI) confirming plantar fasciitis/fasciosis
  * Symptoms consistent with plantar fasciitis/fasciosis for at least 6 months as assessed by patient history
  * Pain unresponsive to non-steroidal anti-inflammatory drugs (NSAIDs) and any four of the following conservative treatments: rest, taping, orthotics, shoe modifications, night splinting, casting, physical therapy, or local corticosteroid injections for up to 3 months
* Must be at least 18 years old and no more than 72 years old
* Must sign the Institutional Review Board (IRB) approved informed consent form
* Subject is willing and able to complete required follow-up

Exclusion Criteria:

* Body mass index (BMI) > 40
* History or documentation showing type I and type II diabetes mellitus
* Physical findings and documentation of coagulopathy, infection, tumor or other systemic disease(s)
* History or documentation showing peripheral vascular disease or autoimmune disease
* Subject has received NSAIDs (e.g., ibuprofen, naproxen) for treatment of plantar fasciitis/fasciosis 2 weeks prior to treatment by this study
* Subject has received NSAIDs (e.g. ibuprofen, naproxen) or oral corticosteroids 2 weeks prior to treatment by this study
* Subject is receiving worker's compensation
* Subject is currently involved in litigation related to the injury being studied
* Prior surgical treatment of the plantar fascia(s) to be treated by this study
* Subject is currently participating in another drug/device study related to the injured plantar fascia
* Pregnant or pregnant suspected subjects
* Clinically significant bilateral plantar fasciitis/fasciosis with a VAS pain scale of > 5 bilaterally
* Subject is not capable of understanding or responding to study questionnaires.
* Extracorporeal shockwave therapy (ESWT) within 6 months of study treatment

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pain relief | at 24 hours, 48 hours, 7 to 14 days, 4 to 6 weeks, 3 months, 6 months, 12 months

SECONDARY OUTCOMES:
Compare the number of postoperative complications | When and if they occur
Evaluate changes in biomechanical function using Ankle-Hindfoot and Midfoot Scale | 4 to 6 weeks, 3 months, 6 months and 1 year
Assess function and quality of life by the sf-36 questionnaire | at 4 to 6 weeks, 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lowell S. Weil, Sr., DPM, Principal Investigator — Weil Foot & Ankle Institute
Locations (1):
- Weil Foot & Ankle Institute, Des Plaines, Illinois, United States